CLINICAL TRIAL: NCT01584687
Title: mRNA Expression as a Biomarker of Xolair (Omalizumab) Response
Brief Title: mRNA Expression as a Biomarker of Omalizumab Response
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Instituto de Investigação em Imunologia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIGE025ABR03T
Record Dates: First submitted 2012-04-20; First posted 2012-04-25 (Estimated); Last update posted 2012-04-25 (Estimated); Status verified 2012-04

CONDITIONS: Asthma
Keywords: asthma; difficult-to-control asthma; mRNA expression; biomarker; real time PCR; ACT; ACQ
MeSH Terms: conditions — Asthma | interventions — Omalizumab; anti-IgE antibodies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Omalizumab (Experimental): All patients will receive omalizumab.
  Interventions: Biological: Omalizumab

INTERVENTIONS:
Biological: Omalizumab — The patients will receive Omalizumab according to their age and weight for 4 months.
  Other Names: Anti-IgE; Xolair

SUMMARY:
Objectives: 1. Determine if mRNA expression could be use as a biomarker to predict and monitor the response to omalizumab in patients with difficult control asthma 2. Identify which genes are switched on and which are switched off by using Omalizumab.

Methods: This study is an open label clinical trial, with six patients. The patients will receive Omalizumab according to their age and weight (maximum dose: 375 mg every 15 days) for 4 months. There will be a run-in period of one month, when allergic asthma diagnosis will be confirmed and treatment will be optimized. Patients will be evaluated and will have blood sample collected on 3 occasions: in the beginning, 2 months after baseline and at the end of the study. Blood samples will always be collected one week after the last omalizumab dose. Primary outcome will be RNA expression of 20 genes measured by real time-PCR (high-affinity IgE receptor, IL-4, IL-5, IL-13, gama-IFN, quimokines, Fc epsilon, between others). Secondary outcomes will be ACT, ACQ and spirometry.

DETAILED DESCRIPTION:
Study rational: There is not a biomarker that can predict which patients will respond to Omalizumab and those who will not respond. Nowadays, the monitoring of therapeutic response to Omalizumab is based on clinical and spirometric data.

On the other hand, when a medication is administered, it has its main expected effect, but also acts on other targets with various direct and indirect effects. We do not know all the genes that are switched on and those that are switched off by the use of Omalizumab. For example, anti-IgE has been developed to block serum total IgE and thereby improve control of allergic asthma. However, the studies noted that Omalizumab also reduces the receptors FcepsilonRI, which may have implications for the treatment of autoimmune urticaria.

ELIGIBILITY:
Inclusion Criteria:

* over 12 years
* severe asthma not controlled despite medication
* IgE between 70 and 1300 IU/ml and evidence of allergy clinical history and/or skin test or blood.

Exclusion Criteria:

* previous use of omalizumab
* smoke history

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Estimated)
Dates: Start 2012-06; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Change of mRNA expression in leukocytes (real time-PCR) | At the end of the study (4months after baseline)
  Patients will be evaluated and will have blood sample collected on 3 occasions: in the beginning, 2 months after baseline and at the end of the study. Blood samples will always be collected one week after the last omalizumab dose. Primary outcome will be RNA expression of 30 genes measured by real time-PCR.

SECONDARY OUTCOMES:
Change in the scores of questionnaires of asthma control | At the end of the study (4 months after baseline)
  Patients will be evaluated on 3 occasions: in the beginning, 2 months after baseline and at the end of the study. Secondary outcomes will be the scores of Asthma Control Test and Asthma Control Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Giavina-Bianchi, MD,PhD, Principal Investigator — University of Sao Paulo